CLINICAL TRIAL: NCT07040462
Title: Child-Parent Psychotherapy for Post-Earthquake Trauma in Preschool Children: A Randomized Controlled Trial
Brief Title: Child-Parent Psychotherapy After the 2023 Kahramanmaraş Earthquake
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beykoz University (Other)
Collaborators: Istanbul Nisantasi University (Other)
Responsible Party: Principal Investigator, Eda Yilmazer, Dr, Beykoz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPP-Kahramanmaras-RCT-2025
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Post-Traumatic Stress Disorder Complex; Emotional Dysregulation
Keywords: Child-Parent Psychotherapy (CPP); Trauma Therapy; Preschool Children; Kahramanmaraş Earthquake

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel arms: (1) Child-Parent Psychotherapy (CPP) or (2) No-treatment control. Each participant remains in their assigned arm throughout the 12-week study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Child-Parent Psychotherapy (CPP) (Experimental): Participants in this arm will receive 12 weekly Child-Parent Psychotherapy (CPP) sessions, each lasting approximately 60 minutes. CPP is a trauma-informed, attachment-based intervention that integrates psychodynamic, cognitive-behavioral, and developmental principles. Sessions are dyadic (child and caregiver together) and may be conducted face-to-face or online. Therapists are trained clinical psychologists. The intervention focuses on emotional regulation, trauma narrative development, and strengthening the caregiver-child bond.
  Interventions: Behavioral: Child-Parent Psychotherapy (CPP)
- No-Treatment Control (No Intervention): Participants in this arm will receive no psychological intervention during the 12-week study period. They will, however, complete outcome assessments at the same three timepoints as the intervention group (baseline, mid-intervention, and post-intervention).

INTERVENTIONS:
Behavioral: Child-Parent Psychotherapy (CPP) — CPP is a structured, evidence-based dyadic therapy designed for children aged 0-6 exposed to trauma and their caregivers. The intervention involves weekly joint sessions emphasizing safety, emotional expression, and caregiver reflective functioning. Delivered by trained psychologists either online or in person.
  Arms: Child-Parent Psychotherapy (CPP)

SUMMARY:
This study aims to evaluate the effectiveness of Child-Parent Psychotherapy (CPP) in reducing trauma-related symptoms and improving attachment quality among preschool-aged children who experienced the 2023 Kahramanmaraş earthquakes in Türkiye. A total of 60 caregiver-child dyads (children aged 3-6) will be recruited from 11 earthquake-affected provinces. Participants will be randomly assigned to either the intervention group, receiving 12 weekly CPP sessions, or a no-intervention control group. CPP will be delivered by trained clinical psychologists through either online or face-to-face sessions. Assessments will be conducted at baseline, mid-intervention (after session 6), and post-intervention (after session 12). Outcomes include child trauma symptoms, social-emotional functioning, and attachment quality, as well as caregiver reflective functioning, stress, and emotional well-being.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the impact of Child-Parent Psychotherapy (CPP) on post-traumatic recovery and attachment in children aged 3 to 6 years who were exposed to the 2023 Kahramanmaraş earthquakes. CPP is a trauma-informed dyadic therapy that integrates psychodynamic, cognitive-behavioral, attachment, and developmental principles, emphasizing co-construction of trauma narratives and caregiver reflective functioning through play-based interaction.

The study will enroll 60 caregiver-child dyads from the 11 most affected cities in Türkiye: Kahramanmaraş, Hatay, Adıyaman, Gaziantep, Malatya, Adana, Osmaniye, Diyarbakır, Şanlıurfa, Kilis, and Elazığ. Eligible participants include children who were between 1-4 years old at the time of the disaster and are currently aged 3-6, along with a primary caregiver (mother or father) who is consistently involved in daily care.

The intervention group will receive 12 weekly CPP sessions (60 minutes each), conducted either online or in person, depending on logistical and contextual needs. Sessions will be delivered by licensed clinical psychologists trained in the CPP protocol. The control group will receive no intervention during the trial period but will complete assessments in parallel with the intervention group.

Primary outcomes include reduction in child trauma symptoms and improvement in social-emotional functioning and attachment quality. Secondary outcomes include parental stress, reflective functioning, and symptoms of depression, anxiety, and stress. Data will be collected at three timepoints: baseline (T1), mid-intervention (after session 6, T2), and post-intervention (after session 12, T3).

All instruments are validated in Turkish populations and age-appropriate. The child measures include the Ages & Stages Questionnaires: Social-Emotional (ASQ:SE), Brief Attachment Scale (BAS-16), and a trauma symptom checklist appropriate for preschoolers. Caregiver measures include the Parental Reflective Functioning Questionnaire (PRFQ), Parenting Stress Index Short Form (PSI-SF), and the Depression Anxiety Stress Scale (DASS-21).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 6 years old at the time of enrollment
* Resided in one of the 11 cities affected by the 2023 Kahramanmaraş earthquake (e.g., Hatay, Kahramanmaraş, Adıyaman, Malatya, Gaziantep, Şanlıurfa, Adana, Osmaniye, Diyarbakır, Kilis, Elazığ)
* Exposure to at least one qualifying traumatic event due to the earthquake (e.g., witnessing injury or death, loss of home, separation from caregiver)
* Living with a primary caregiver (mother or father) who consents to participate in the study
* Both caregiver and child are available to participate in 12 weekly sessions of CPP (online or face-to-face)
* Caregiver is fluent in Turkish and able to complete self-report questionnaires

Exclusion Criteria:

* Child or caregiver currently receiving psychotherapy or psychiatric treatment
* Child diagnosed with developmental disorder (e.g., autism, intellectual disability) that significantly impairs communication or relational functioning
* Caregiver with a diagnosed severe psychiatric disorder (e.g., psychosis, bipolar disorder) or active substance use disorder
* Families with ongoing legal custody disputes or instability that may interfere with consistent participation
* Inability to access internet or digital device (for participants randomized to online therapy)

Ages: 3 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in Child Trauma Symptom Severity | From baseline (Week 0) to 12 weeks post-intervention.
  Child trauma symptoms will be assessed using the Child PTSD Reaction Index (CPTSD-RI), a 20-item caregiver-report scale developed to evaluate post-traumatic stress reactions in children following exposure to traumatic events. Items are rated on a 5-point Likert scale ranging from 0 (none) to 4 (most of the time), yielding a total score ranging from 0 to 80. Higher scores reflect greater severity of PTSD symptoms, with cutoffs indicating doubtful (0-11), mild (12-24), moderate (25-39), severe (40-59), and very severe (60-80) symptom levels. The measure will be administered at three time points: baseline (Week 0), mid-treatment (Week 6), and post-treatment (Week 12).

SECONDARY OUTCOMES:
Change in Child Social-Emotional Functioning | From baseline (Week 0) to 12 weeks post-intervention.
  Assessed using the ASQ:SE, a caregiver-report scale evaluating emotion regulation, social interaction, and adaptive functioning. Total scores vary by age version, typically up to ~310. Higher scores indicate more social-emotional difficulties.
Change in Child Attachment Security | From baseline (Week 0) to 12 weeks post-intervention.
  Measured using the BAS-16, a 16-item scale assessing attachment security and proximity-seeking. Scores range from 16 to 80, with higher scores indicating more secure attachment.
Change in Parental Reflective Functioning | From baseline (Week 0) to 12 weeks post-intervention.
  Evaluated using the PRFQ, an 18-item caregiver-report measure of mentalization. Scores range from 18 to 126, with interpretation based on subscale balance.
Change in Parenting Stress | From baseline (Week 0) to 12 weeks post-intervention
  Measured by the PSI-SF, a 36-item scale with scores ranging from 36 to 180, where higher scores indicate greater stress.
Change in Caregiver Depression, Anxiety, and Stress | From baseline (Week 0) to 12 weeks post-intervention.
  Assessed by the DASS-21, which yields three subscale scores (each 0-42) for depression, anxiety, and stress. Higher scores indicate greater emotional distress.

CONTACTS AND LOCATIONS:
Locations (1):
- Beykoz University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in this study (after de-identification) will be made available to researchers who provide a methodologically sound proposal. Data will include participant-level data for primary and secondary outcomes. Supporting documents such as the study protocol, statistical analysis plan, and informed consent form will also be made available upon request. Data will be available beginning 6 months after publication of the main findings and will remain accessible for 3 years via a secure institutional repository or upon request to the principal investigator.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available 6 months after publication of the study results and remain accessible for 5 years.
Access Criteria: Requests should be submitted to the principal investigator and will be evaluated based on the scientific validity and ethical compliance of the proposal.